CLINICAL TRIAL: NCT03591887
Title: A Phase II, Randomized, Parallel Group, Placebo-controlled, Double-blinded, Dose-finding Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of ABY-035 in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Study to Evaluate ABY-035 in Subjects With Moderate-to-severe Plaque Psoriasis
Acronym: AFFIRM-35
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affibody (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABY-035-002; 2017-001615-36 (EudraCT Number)
Record Dates: First submitted 2018-06-01; First posted 2018-07-19 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ABY-035 2 mg (Experimental): 2 mg ABY-035 SC
  Interventions: Biological: ABY-035
- ABY-035 20 mg (Experimental): 20 mg ABY-035 SC
  Interventions: Biological: ABY-035
- ABY-035 80 mg (Experimental): 80 mg ABY-035 SC
  Interventions: Biological: ABY-035
- ABY-035 160 mg (Experimental): 160 mg ABY-035 SC
  Interventions: Biological: ABY-035
- Placebo (Placebo Comparator): Placebo, switching to 80 mg ABY-035 after 12 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ABY-035 — ABY-035 solution for injection
  Arms: ABY-035 160 mg; ABY-035 2 mg; ABY-035 20 mg; ABY-035 80 mg
Biological: Placebo — Placebo to ABY-035 solution for injection
  Arms: Placebo

SUMMARY:
This randomized, double-blinded dose-finding study evaluates four dose levels of ABY-035, in comparison to placebo, in subjects with moderate to severe plaque psoriasis.

The study consists of 52-week Core study and two optional 52-week periods, Extension and Prolongation of Extension.

The Core study consists of three periods: Induction (placebo-controlled, Week 0-12), Optimization (Week 12-24), and Individualization (Week 24-52).

DETAILED DESCRIPTION:
The Core study evaluates four doses of ABY-035, in comparison to placebo, in subjects with moderate to severe plaque psoriasis. The treatment periods in the Core study are:

* Induction (Week 0-12) - four dose levels and placebo (Q2W)
* Optimization (Week 12-24) - starting with a possible dose adjustment (all subjects on Q2W) depending on PASI score. Subjects on placebo switch to active drug (Q4W).
* Individualization (Week 24-52) - starting with a switch to Q4W for all subjects. From week 32 dosing interval alters depending on PASI score.

The study is unblinded after completion of the Core study. During the optional Extension and Prolongation of Extension periods, dose levels and intervals alter depending on PASI score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with plaque psoriasis of at least 6 months prior to Screening, without clinically significant flares during the 12 weeks before randomization, with or without psoriatic arthritis
* Having precedent failure, intolerance and/or contraindication to at least two standard therapies for moderate to-severe plaque psoriasis (systemic therapy and/or phototherapy), and previousinsufficient disease control of topical therapy (e.g. corticosteroids, vitamin D derivatives, cignolin/dithranol).
* Moderate-to-severe plaque psoriasis at Screening and at Baseline as defined by:

  i. Psoriasis involving ≥10% BSA ii. PASI score of ≥ 12 iii. sPGA score of ≥ 3
* Use of highly effective method of contraception or female of non-childbearing potential

Exclusion Criteria:

* Current forms of psoriasis other than chronic plaque-type
* Current drug induced psoriasis
* History of hypersensitivity or allergy to the IMP or its excipients
* History of recurrent or medically important infections requiring intervention and/or systemic treatment in the last 12 months, including infections with e.g. candida and Staphylococcus aureus
* History of or any signs of lymphoproliferative disease, or a known malignancy or a history of malignancy within the previous 5 years (with the exception of basal cell or squamous cell carcinoma of the skin that had been fully excised with no evidence of recurrence)
* Autoimmune disease of relevance
* Inflammatory Bowel Disease requiring treatment within the past 12 months
* Clinically significant heart condition which is not well controlled by current therapy, as assessed by the Investigator
* Significantly immunocompromised subject
* Blood pressure out of range
* Laboratory values out of range, including ALT, AST, eGFR
* Positive to HIV, hepatitis B, hepatitis C or tuberculosis
* Recent previous psoriasis treatments, within defined wash-out periods
* Prior exposure to systemic psoriasis treatments with anti-IL-17 biological therapies
* Live vaccination within defined time restrictions
* Inability or unwillingness to limit ultraviolet (UV) light exposure during the course of the study
* Pregnancy, breast feeding
* Drug and/or alcohol abuse or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a ≥90% improvement in Psoriasis Area and Severity Index (PASI90) at week 12 | 12 weeks
  The PASI combines the extent of body surface involvement in the body regions head, trunk, arms, and legs. The percent area of the skin involved is estimated per region (0-100%). The severity is estimated by clinical signs of erythema, induration and scaling, from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Overall scores range from 0 (no psoriasis) to 72 (the most severe disease). PASI90 is a ≥90% reduction from Baseline in PASI score

SECONDARY OUTCOMES:
Number of treatment emergent Adverse Events | 52 weeks
  Adverse Events starting after first administration of study drug
Proportion of subjects achieving a ≥90% improvement in PASI (PASI90) at week 24 | 24 weeks
  A ≥90% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥90% improvement in PASI (PASI90) at week 52 | 52 weeks
  A ≥90% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥50% improvement in PASI (PASI50) at week 12 | 12 weeks
  A ≥50% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥50% improvement in PASI (PASI50) at week 24 | 24 weeks
  A ≥50% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥50% improvement in PASI (PASI50) at week 52 | 52 weeks
  A ≥50% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥75% improvement in PASI (PASI75) at week 12 | 12 weeks
  A ≥75% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥75% improvement in PASI (PASI75) at week 24 | 24 weeks
  A ≥75% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥75% improvement in PASI (PASI75) at week 52 | 52 weeks
  A ≥75% reduction from Baseline in PASI score
Proportion of subjects achieving a 100% improvement in PASI (PASI100) at week 12 | 12 weeks
  A 100% reduction from Baseline in PASI score
Proportion of subjects achieving a 100% improvement in PASI (PASI100) at week 24 | 24 weeks
  A 100% reduction from Baseline in PASI score
Proportion of subjects achieving a 100% improvement in PASI (PASI100) at week 52 | 52 weeks
  A 100% reduction from Baseline in PASI score
Change from baseline in PASI score at week 12 | Week 12
  PASI: Psoriasis Area and Severity Index
Change from baseline in PASI score at week 24 | Week 24
  PASI: Psoriasis Area and Severity Index
Change from baseline in PASI score at week 52 | Week 52
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving an absolute PASI score ≤1 at week 12 | 12 weeks
  PASI ≤1 equals clear or almost clear skin
Proportion of subjects achieving an absolute PASI score ≤1 at week 24 | 24 weeks
  PASI ≤1 equals clear or almost clear skin
Proportion of subjects achieving an absolute PASI score ≤1 at week 52 | 52 weeks
  PASI ≤1 equals clear or almost clear skin
Proportion of subjects achieving an absolute PASI score <3 at week 12 | 12 weeks
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving an absolute PASI score <3 at week 24 | 24 weeks
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving an absolute PASI score <3 at week 52 | 52 weeks
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving Static Physician's Global Assessment (sPGA) 1 or 0 at week 12 | 12 weeks
  The sPGA is the physician's determination of the subject's Psoriasis lesions overall at a given time point, with the grading 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe)
Proportion of subjects achieving Static Physician's Global Assessment (sPGA) 1 or 0 at week 24 | 24 weeks
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving Static Physician's Global Assessment (sPGA) 1 or 0 at week 52 | 52 weeks
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving ≥2 point improvement from baseline in sPGA at week 12 | 12 weeks
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving ≥2 point improvement from baseline in sPGA at week 24 | 24 weeks
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving ≥2 point improvement from baseline in sPGA at week 52 | 52 weeks
  sPGA: Static Physician's Global Assessment
Change from baseline in sPGA at week 12 | 12 weeks
  sPGA: Static Physician's Global Assessment
Change from baseline in sPGA at week 24 | 24 weeks
  sPGA: Static Physician's Global Assessment
Change from baseline in sPGA at week 52 | 52 weeks
  sPGA: Static Physician's Global Assessment
Change from baseline in target nail Nail Psoriasis Severity Index (NAPSI) at week 12 | Week 12
  The NAPSI scale is used to evaluate the severity of psoriasis in the fingernail bed and matrix. The nail is divided into quadrants. Each quadrant is given the score 0 (absence) or 1 (presence) for psoriasis in the beds and matrix, respectively. The NAPSI score of a nail is the sum of each quadrant. The maximum score per nail is 8.
  In the target nail NAPSI, the worst affected nail at Baseline is evaluated throughout the study.
Change from baseline in target nail NAPSI at week 24 | Week 24
  NAPSI: Nail Psoriasis Severity Index
Change from baseline in target nail NAPSI at week 52 | Week 52
  NAPSI: Nail Psoriasis Severity Index
Proportion of subjects achieving Dermatology Life Quality Index (DLQI) of 0 or 1 at week 12 | Week 12
  DLQI is a 10-question quality-of-life questionnaire completed by the subject. It covers 6 the domains symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The total scores range from 0 to 30, with higher score indicating greater quality of life impairment.
Proportion of subjects achieving DLQI of 0 or 1 at week 24 | Week 24
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of 0 or 1 at week 52 | Week 52
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of ≤ 5 at Week 12 | Week 12
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of ≤ 5 at Week 24 | Week 24
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of ≤ 5 at Week 52 | Week 52
  DLQI: Dermatology Life Quality Index
Change from baseline in DLQI at week 12 | Week 12
  DLQI: Dermatology Life Quality Index
DLQI at week 24 compared to baseline | Week 24
  DLQI: Dermatology Life Quality Index
DLQI at week 52 compared to baseline | Week 52
  DLQI: Dermatology Life Quality Index
Change from baseline in pain-Visual Analogue Scale (VAS) at week 12 | Week 12
  Pain-VAS: A patient measurement of level pain, from 0 (no pain) to 100 (worst possible pain)
Pain-VAS score at Week 24 compared to baseline | Week 24
  Pain-VAS: A patient measurement of level pain, from 0 (no pain) to 100 (worst possible pain)
Pain-VAS score at Week 52 compared to baseline | Week 52
  Pain-VAS: A patient measurement of level pain, from 0 (no pain) to 100 (worst possible pain)
Change from baseline in itch-Visual Analogue Scale (VAS) at week 12 | Week 12
  Itch-VAS: A patient measurement of level itching from 0 (no itch) to 100 (worst possible itch)
Itch-VAS at week 24 compared to baseline | Week 24
  Itch-VAS: A patient measurement of level itching from 0 (no itch) to 100 (worst possible itch)
Itch-VAS at week 52 compared to baseline | Week 52
  Itch-VAS: A patient measurement of level itching from 0 (no itch) to 100 (worst possible itch)
Pharmacokinetics: Area Under the Curve (AUC) of ABY-035 | 52 weeks
  AUC is a measure of the drug exposure
Levels of anti-ABY-035 antibodies in serum | 52 weeks
  Anti-drug antibodies
Number of treatment emerging Adverse Events during the Extension period | Week 52 to Week 104
  Adverse Events starting after first administration of study drug
Number of treatment emerging Adverse Events during the Prolongation of Extension period | Week 104 to Week 156
  Adverse Events starting after first administration of study drug
Pharmacokinetics: Area Under the Curve (AUC) of ABY-035 during the Extension period | Week 52 to Week 104
  AUC is a measure of the drug exposure
Pharmacokinetics: Area Under the Curve (AUC) of ABY-035 during the Prolongation of Extension period | Week 104 to Week 156
  AUC is a measure of the drug exposure
Levels of anti-ABY-035 antibodies in serum during the Extension period | Week 52 to Week 104
  Anti-drug antibodies
Levels of anti-ABY-035 antibodies in serum during the Prolongation of Extension period | Week 104 to Week 156
  Anti-drug antibodies
Proportion of subjects achieving a ≥90% improvement in PASI (PASI90) at end of Extension period | Week 104
  A ≥90% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥90% improvement in PASI (PASI90) at end of Prolongation of Extension period | Week 156
  A ≥90% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥50% improvement in PASI (PASI50) at end of Extension period | Week 104
  A ≥50% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥50% improvement in PASI (PASI50) at end of Prolongation of Extension period | Week 156
  A ≥50% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥75% improvement in PASI (PASI75) at end of Extension period | Week 104
  A ≥75% reduction from Baseline in PASI score
Proportion of subjects achieving a ≥75% improvement in PASI (PASI75) at end of Prolongation of Extension period | Week 156
  A ≥75% reduction from Baseline in PASI score
Proportion of subjects achieving a 100% improvement in PASI (PASI100) at end of Extension period | Week 104
  A 100% reduction from Baseline in PASI score
Proportion of subjects achieving a 100% improvement in PASI (PASI100) at end of Prolongation of Extension period | Week 156
  A 100% reduction from Baseline in PASI score
Change from baseline in PASI score at end of Extension period | Week 104
  PASI: Psoriasis Area and Severity Index
Change from baseline in PASI score at end of Prolongation of Extension period | Week 156
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving an absolute PASI score ≤1 at end of Extension period | Week 104
  PASI ≤1 equals clear or almost clear skin
Proportion of subjects achieving an absolute PASI score ≤1 at end of Prolongation of Extension period | Week 156
  PASI ≤1 equals clear or almost clear skin
Proportion of subjects achieving an absolute PASI score <3 at end of Extension period | Week 104
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving an absolute PASI score <3 at end of Prolongation of Extension period | Week 156
  PASI: Psoriasis Area and Severity Index
Proportion of subjects achieving sPGA of 0 or 1 at end of Extension period | Week 104
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving sPGA of 0 or 1 at end of Prolongation of Extension period | Week 156
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving ≥2 point improvement from baseline in sPGA at end of Extension period | Week 104
  sPGA: Static Physician's Global Assessment
Proportion of subjects achieving ≥2 point improvement from baseline in sPGA at end of Prolongation of Extension period | Week 156
  sPGA: Static Physician's Global Assessment
Change from baseline in sPGA at end of Extension period | Week 104
  sPGA: Static Physician's Global Assessment
Change from baseline in sPGA at end of Prolongation Extension period | Week 156
  sPGA: Static Physician's Global Assessment
Change from baseline in target nail NAPSI at end of Extension period | Week 104
  NAPSI: Nail Psoriasis Severity Index
Change from baseline in target nail NAPSI at end of Prolongation of Extension period | Week 156
  NAPSI: Nail Psoriasis Severity Index
Proportion of subjects achieving DLQI of 0 or 1 at end of Extension period | Week 104
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of 0 or 1 at end of Prolongation of Extension period | Week 156
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of ≤ 5 at end of Extension period | Week 104
  DLQI: Dermatology Life Quality Index
Proportion of subjects achieving DLQI of ≤ 5 at end of Prolongation of Extension period | Week 156
  DLQI: Dermatology Life Quality Index
DLQI at end of Extension period compared to baseline | Week 104
  DLQI: Dermatology Life Quality Index
DLQI at end of Prolongation of Extension period compared to baseline | Week 156
  DLQI: Dermatology Life Quality Index
Pain-VAS score at end of Extension period compared to baseline | Week 104
  Pain-VAS: A patient measurement of level pain, from 0 (no pain) to 100 (worst possible pain)
Pain-VAS at end of Prolongation of Extension period compared to baseline | Week 156
  Pain-VAS: A patient measurement of level pain, from 0 (no pain) to 100 (worst possible pain)
Itch-VAS at end of Extension period compared to baseline | Week 104
  Itch-VAS: A patient measurement of level itching from 0 (no itch) to 100 (worst possible itch)
Itch-VAS at end of Prolongation of Extension period compared to baseline | Week 156
  Itch-VAS: A patient measurement of level itching from 0 (no itch) to 100 (worst possible itch)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Gerdes, Dr. med, Principal Investigator — Klinik für Dermatologie, Venerologie und Allergologie
Locations (18):
- Germany (18):
  - Rothhaar Studien GmbH, Berlin
  - Praxis für Haut- und Geschlechtskrankheiten im Ärztehaus "Rudolf Virchow", Berlin
  - Hautzentrum Weissensee, Berlin
  - Hautarztzentrum Tegel, Berlin
  - Klinik für Dermatologie, Venerologie und Allergologie der Ruhr-Universität, Bochum
  - Hautarztpraxis im Jahrhunderthaus, Bochum
  - RuhrDerm - Studienzentrum der Gemeinschaftspraxis für Dermatologie, Venerologie, Allergologie, Phlebologie, Bochum
  - Elbe Kliniken Buxtehude, Buxtehude
  - Rosenpark Research, Darmstadt
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Derma-Study-Center FN GmbH, Friedrichshafen
  - SCIderm Clinics, Hamburg
  - Klinik für Dermatologie, Venerologie und Allergologie, Kiel
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Clinical research center (CRC) Department of Dermatology, Mainz
  - Dres. Unnewehr, Osnabrück
  - CMS³ - Company for Medical Study & Service Selters UG, Selters
  - CentroDerm GmbH, Wuppertal

IPD SHARING:
Plan to Share IPD: No